CLINICAL TRIAL: NCT01232491
Title: A 26-week Randomised, Controlled, Open Label, Multicentre, Multinational, Treat to Target Trial Investigating the Impact of Dietary Intervention on Weight Change and the Relationship Between Weight Change and Baseline Body Mass Index (BMI) in Subjects With Type 2 Diabetes Inadequately Controlled on Oral Antidiabetic Drugs (OADs) Initiating Insulin Therapy With Insulin Detemir in Combination With Metformin (Levemir DIET)
Brief Title: Impact of Dietary Intervention on Weight Change in Subjects With Type 2 Diabetes
Acronym: DIET™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-3785; U1111-1116-2629 (Other: WHO); 2009-014894-42 (EudraCT Number)
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Insulin detemir (Levemir®) 100 U/mL, was injected subcutaneously once daily with the evening meal or at bedtime as add-on to subject's pre-trial treatment of metformin for 26 weeks. Subjects did not receive dietary consultation except for basic dietary advice at baseline. Insulin doses were individually adjusted.
  Interventions: Drug: Insulin detemir
- Dietician (Experimental): Insulin detemir (Levemir®) 100 U/mL, was injected subcutaneously once daily with the evening meal or at bedtime as add-on to subject's pre-trial treatment of metformin for 26 weeks. Subjects received dietary consultation according to local standard during 3 face-to-face meetings and 3 phone contacts. Insulin doses were individually adjusted.
  Interventions: Drug: Insulin detemir; Dietary Supplement: Dietary regimen

INTERVENTIONS:
Drug: Insulin detemir — Individually adjusted insulin detemir subcutaneously (under the skin) once daily. Subjects continue their pre-trial metformin treatment.
Dietary Supplement: Dietary regimen — Subjects receive dietary consultation by a dietician at six occasions during the trial.
  Arms: Dietician

SUMMARY:
This trial is conducted in Europe, and North and South America. The aim of this trial is to investigate if a dietary intervention has an effect on weight when initiating insulin treatment in subjects with type 2 diabetes currently treated with oral antidiabetic drugs (OADs).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (diagnosed clinically) for at least 6 months prior trial start
* Insulin naive subjects
* HbA1c: 7.0-9.0 % (both inclusive)
* Body Mass Index (BMI): 25.0-45.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Use of Thiazolidinedione (TZDs) or Glucagon-like peptide-1 analogue (GLP- 1) receptor agonists within the last 3 months prior to trial enrollment
* Cardiovascular disease within the last 6 months
* Recurrent severe hypoglycaemia or hypoglycaemic unawareness or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Uncontrolled treated/untreated severe hypertension, impaired liver function, impaired renal function, known proliferative retinopathy or maculopathy requiring treatment
* Cancer and medical history of cancer in the past 5 years (except basal cell skin cancer or squamous cell skin cancer)
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2010-10-29 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2011-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry Gorsøe (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (97):
- United States (66):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Ozark, Alabama
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Burlingame, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, National City, California
  - Novo Nordisk Investigational Site, Redlands, California
  - Novo Nordisk Investigational Site, Santa Ana, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Norwalk, Connecticut
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Jupiter, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Perry, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Oympiafields, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Shawnee Mission, Kansas
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Portland, Maine
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Brockton, Massachusetts
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Southfield, Michigan
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Durham, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Jenkintown, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Anderson, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Rapid City, South Dakota
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Odessa, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Martinsburg, West Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Argentina (5):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Caba
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Godoy Cruz
- Germany (7):
  - Novo Nordisk Investigational Site, Bad Neuenahr-Ahrweiler
  - Novo Nordisk Investigational Site, Gelnhausen
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Marburg
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Völklingen
- Poland (4):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Torun
  - Novo Nordisk Investigational Site, Warsaw
- Puerto Rico (2):
  - Novo Nordisk Investigational Site, Carolina
  - Novo Nordisk Investigational Site, Manatí
- Novo Nordisk Investigational Site, Saint Petersburg, Russia
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Slovakia (3):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Ľubochňa
- Slovenia (3):
  - Novo Nordisk Investigational Site, Koper
  - Novo Nordisk Investigational Site, Maribor
  - Novo Nordisk Investigational Site, Novo Mesto
- Spain (2):
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Sanlúcar de Barrameda
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Samsun

REFERENCES:
- [Background] Niswender K, Piletic M, Andersen H, Conradsen Hiort L, Hollander P. Weight change upon once-daily initiation of insulin detemir with or without dietary intervention in overweight or obese insulin-naive individuals with type 2 diabetes: results from the DIET trial. Diabetes Obes Metab. 2014 Feb;16(2):186-92. doi: 10.1111/dom.12218. Epub 2013 Oct 29. PMID 24112375
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 110 sites in 9 countries: Argentina (5), Germany (7), Poland (4), Serbia (4), Slovakia (3), Slovenia (2), Spain (4), Turkey (5) and United States of America (76).
Pre-assignment Details: Subjects continued on their treatment with metformin, at the pre-randomisation dose level and dosing frequency. All other oral antidiabetic drugs were discontinued before insulin detemir was used.
Period: Overall Study
Arm/Group | Dietician | Control
Started | 306 | 305
Exposed (Safety Analysis Set) | 305 (One subject withdrew prior to exposure to trial drug.) | 301 (Four subjects withdrew prior to exposure to trial drug.)
Completed | 246 | 242
Not Completed | 60 | 63
Not completed — Adverse Event | 13 | 8
Not completed — Lack of Efficacy | 1 | 5
Not completed — Protocol Violation | 13 | 11
Not completed — Withdrawal Criteria | 12 | 21
Not completed — Other | 21 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dietician | Control | Total
Number analyzed (Participants) | 305 | 301 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.7) | 56.5 (10.0) | 57.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 143 | 295
  Male | 153 | 158 | 311
Race/Ethnicity, Customized [Number; unit: participants]
  White | 274 | 268 | 542
  Black or African American | 21 | 26 | 47
  Asian | 2 | 5 | 7
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Oth. Pacific Islander | 3 | 0 | 3
  Other | 5 | 2 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 63 | 78 | 141
  Not Hispanic or Latino | 242 | 223 | 465
Height [Mean (Standard Deviation); unit: meters] | 1.67 (0.10) | 1.68 (0.10) | 1.67 (0.10)
Body weight [Mean (Standard Deviation); unit: kg] | 96.4 (18.2) | 97.0 (20.4) | 96.7 (19.3)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.4 (5.4) | 34.3 (5.6) | 34.4 (5.5)
Duration of diabetes [Mean (Standard Deviation); unit: years] — The number of subjects (N) analysed in the Dietician group was 303 instead of 305.
  years | 8.6 (5.8) | 8.5 (6.0) | 8.6 (5.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — The number of subjects (N) analysed in the Control group was 298 instead of 301.
  mmol/L | 9.3 (2.3) | 9.2 (2.0) | 9.2 (2.2)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.0 (0.7) | 7.9 (0.6) | 7.9 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Weight
Description: Estimated mean change from baseline in body weight after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects and missing data is imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Dietician | Control
Number analyzed (Participants) | 306 | 305
kg | -1.05 (0.23) | -0.56 (0.23)
Statistical Analysis 1: Comparison: Dietician vs Control; Normal linear regression model with treatment, strata, use of insulin secretagogue at screening, sex and region as factors and age and weight at baseline as covariates. Superiority was considered confirmed if the upper bound of the two-sided 95% CI for the estimated treatment difference (dietary intervention versus no dietary intervention), which was calculated using the FAS, was below 0 kg; Test type: Superiority or Other; p = 0.132, Regression, Linear — If the p-value for the two-sided test was less than 5%, and D (the estimated treatment difference [dietary intervention versus no dietary intervention]) was less than 0 then superiority for dietary intervention was considered confirmed; Estimated treatment difference, LS Mean = 0.49, 95% CI [-0.15 to 1.13]

2. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Estimated mean change from baseline in BMI after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Dietician | Control
Number analyzed (Participants) | 306 | 305
kg/m^2 | -0.37 (0.08) | -0.20 (0.08)
Statistical Analysis 1: Comparison: Dietician vs Control; Normal linear regression model with treatment, use of insulin secretagogue at screening, sex and region as factors, and age and BMI at baseline as covariates; Test type: Superiority or Other; p = 0.137, Regression, Linear; Estimated treatment difference, LS Mean = 0.17, 95% CI [-0.05 to 0.39]

3. Secondary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c)
Description: Estimated mean change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Dietician | Control
Number analyzed (Participants) | 306 | 305
percentage of glycosylated haemoglobin | -0.93 (0.05) | -0.80 (0.05)
Statistical Analysis 1: Comparison: Dietician vs Control; Normal linear regression model with treatment, strata, use of insulin secretagogue at screening and region as factors and HbA1c at baseline as covariate; Test type: Superiority or Other; p = 0.053, Regression, Linear; Estimated treatment difference, LS Mean = 0.13, 95% CI [-0.00 to 0.26]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Estimated mean change from baseline in FPG after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Dietician | Control
Number analyzed (Participants) | 306 | 302
mmol/L | -3.00 (0.12) | -2.93 (0.12)
Statistical Analysis 1: Comparison: Dietician vs Control; Normal linear regression model with treatment, strata, use of insulin secretagogue at screening and region as factors and FPG at baseline as covariate; Test type: Superiority or Other; p = 0.674, Regression, Linear; Estimated treatment difference, LS Mean = 0.07, 95% CI [-0.25 to 0.39]

5. Secondary Outcome: Rate of Treatment Emergent Adverse Events (TEAEs)
Description: Corresponds to rate of adverse events (AEs) per 100 patient years of exposure. Mild AEs: no or transient symptoms, no interference with subject's daily activities. Moderate AEs: marked symptoms, moderate interference with subject's daily activities. Severe AEs: considerable interference with subject's daily activities, unacceptable. Serious AEs: AEs that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalization, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 26
Population: Safety analysis set includes all subjects who received at least one dose of insulin detemir.
Measure: Number; unit: rate per 100 years of patient exposure
Arm/Group | Dietician | Control
Number analyzed (Participants) | 305 | 301
rate per 100 years of patient exposure
  All TEAEs | 387.9 | 437.1
  Serious TEAEs | 16.3 | 16.6
  Severe TEAEs | 16.3 | 11.3
  Moderate TEAEs | 130.5 | 108.3
  Mild TEAEs | 241.0 | 317.5

6. Secondary Outcome: Rate of All Treatment Emergent Hypoglycaemic Episodes
Description: Corresponds to rate of treatment emergent hypoglycaemic episodes per patient exposure year. A hypoglycaemic episode was defined as treatment emergent if the onset of the episode was on or after the first day of exposure to randomised treatment and no later than 1 day after the last day of randomised treatment. Severe, if assistance was required to actively administer carbohydrate, glucagons or other resuscitative actions.
Time Frame: Week 0 to Week 26
Population: Safety analysis set includes all subjects who received at least one dose of insulin detemir.
Measure: Number; unit: rate per year of patient exposure
Arm/Group | Dietician | Control
Number analyzed (Participants) | 305 | 301
rate per year of patient exposure
  All Events | 25.47 | 23.30
  Severe Events | 0.01 | 0.01

7. Secondary Outcome: Rate of Nocturnal Treatment Emergent Hypoglycaemic Episodes
Description: Corresponds to rate of treatment emergent hypoglycaemic episodes per patient exposure year. A hypoglycaemic episode was defined as treatment emergent if the onset of the episode was on or after the first day of exposure to randomised treatment and no later than 1 day after the last day of randomised treatment. A hypoglycaemic episode with time of onset between 00:01 and 05:59 a.m. (both included) was considered nocturnal. Severe, if assistance was required to actively administer carbohydrate, glucagons or other resuscitative actions.
Time Frame: Week 0 to Week 26
Population: Safety analysis set includes all subjects who received at least one dose of insulin detemir.
Measure: Number; unit: rate per year of patient exposure
Arm/Group | Dietician | Control
Number analyzed (Participants) | 305 | 301
rate per year of patient exposure
  All Events | 5.59 | 5.51
  Severe Events | 0.01 | 0.01

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks.
Description: Safety analysis set includes all subjects who received at least one dose of insulin detemir.
Arm/Group | Dietician | Control
Serious Adverse Events (participants affected / at risk) | 17/305 | 19/301
Other Adverse Events (participants affected / at risk) | 61/305 | 69/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietician (N=305) | Control (N=301)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (3) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietician (N=305) | Control (N=301)
Injection site reaction (General disorders) | 16 (21) | 13 (17)
Nasopharyngitis (Infections and infestations) | 30 (39) | 38 (49)
Headache (Nervous system disorders) | 23 (29) | 24 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.